CLINICAL TRIAL: NCT04065178
Title: Day-time Activity Level In Inpatient Neurological Rehabilitation as Related to Functional Outcomes at Discharge, Length of Stay, Discharge Location, and Quality of Life: A Preliminary Study
Brief Title: Day Time Activity Level in Inpatient Neurological Rehabilitation as Related to Functional Outcomes at Discharge, Length of Stay, Discharge Location, and Quality of Life: a Preliminary Study
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1050469
Record Dates: First submitted 2019-01-23; First posted 2019-08-22 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Activity Level

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Level of Activity: Level of activity for all patients admitting to the inpatient neurological rehabilitation unit.
  Interventions: Behavioral: Level of activity

INTERVENTIONS:
Behavioral: Level of activity — Inpatients will be asked if they are willing to wear a heart rate tracking fitness watch during their stay. They will be asked quality of life questions on a questionnaire that will take approximately 30 minutes to answer at admission and discharge. At the end of the study they will return the Fitbit Charge 2 to the study coordinator or their nurse.
  Your rehabilitation plan of care will not change in any other way.

SUMMARY:
This preliminary study is intended to collect activity level data in a preliminary longitudinal means in order to gain more knowledge into our patient's current activity status. Our long-term objective of tracking patient activity levels in relation to function and length of stay is to identify opportunities for improved patient activity level, decreased length of stay, and increased functional mobility at discharge.

The main purpose of this study is the exploration of the ability to generate meaningful activity data. Usual standard of care will be taking place during this preliminary study, there is not an intervention being studied at this time.

DETAILED DESCRIPTION:
Identified possible subjects will be approached for Consent to participate by the Study coordinator. Subjects who have previously completed the study, and are re-admitted can be approached for participate if they meet eligibility. If the subject consent is approved, the subject is given a research number that will correlate to their name on a list locked in a separate location by the study coordinator.

The Study coordinator will issue a Fitbit Charge 2 watch for heart rate tracking purposes. The study coordinator will fit the subject with the watch ensuring proper fitting on the non-affected wrist in the event of hemiparesis of the patient in order to collect appropriate movement data and have decreased risk for skin breakdown due to possible impaired sensation on the paretic side. Tests and measures are the same for all patients on the rehab unit and will not vary based on participation in the study. The research coordinator will gather tests and measures performed by clinical staff and compile the data in an organized manner. The research coordinator will amass data in Redcap with tests and measure scores aligned with the subject number. This site is password protected and only available to delegated research staff. The most detailed data collection will be with the wearable heart rate monitoring Fitbit Charge 2 devices.

The device will require battery recharge approximately every 3-5 days, during this time data will also be downloaded. The Fitbit Charge 2 has a charging time of 2 hours, therefore every 3-5 days there will be an approx. 2-3 hour missing data piece during charging and downloading time, charging days will be compared with all other non-charging days to average data. It is acceptable for there to be up to 48 hours of missing data, in which charging and downloading data will take place as well as any procedures the subject may need that would require the Fitbit Charge 2 to be removed. Each subject will have a watch designated to them and each device will have a separate profile within the Fitbit Charge 2 dashboard. Data will be downloaded from the Fitbit Charge 2 dashboard to excel formatting. Profiles of each patient will not include protected health information and profiles will be set up using subject number, birth year, gender, height and weight in order to obtain accurate health metrics. Encrypted data will be stored in the Redcap system.

Fitbit Charge 2 files will be downloaded weekly (every 3-5 days) utilizing .csv file format in summary array. Included metrics are minutes sedentary, minutes lightly active, minutes fairly active, minutes very active, minutes asleep, minutes awake, and time in bed. The research coordinator will keep the timestamp array data for the .csv files organized in Redcap.

Rehab processes will not change based on participation in the study. Within 24 hours of discharge the study coordinator will re-administer the SF-36 quality of life measure, collect equipment, thank the subjects for participation, and assess for any skin breakdown related to the usage of the watch, if not previously done within 24 hours. The study coordinator will ensure data subset is organized and properly stored for the statistician including Fitbit Charge 2 and functional mobility measures.

ELIGIBILITY:
Inclusion criteria:

* English as a first speaking language
* willingness to participate (family consent if patient is not able to consent)
* ability to wear a heart rate tracking device during full admission
* intact skin integrity of the arms
* commercial insurance or government insurance (medicare or medicaid)
* an estimated length of stay greater than 5 days and less than 5 weeks at initial assessment by the admitting team

Exclusion criteria:

* patients with multiple sclerosis (MS), brain tumors, or degenerative neurological disorders
* patients with a pacemaker, left ventricular assist device, or with ventilator support
* patients without health insurance in place
* non-primary English speaking
* patients who require 1:1 supervision as they are deemed unable to comply with device wearing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitting to the Inpatient Neurological Specialty Unit (a rehab unit)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Sedentary Minutes | Length of stay in the inpatient facility-will differ for each patient (expected average of 3 weeks)
  Sedentary minutes will be reported from the Fitbit Charge 2.
Lightly Active Minutes | Length of stay in the inpatient facility-will differ for each patient (expected average of 3 weeks)
  Lightly active minutes will be reported from the Fitbit Charge 2.
Fairly Active Minutes | Length of stay in the inpatient facility-will differ for each patient (expected average of 3 weeks)
  Fairly active minutes will be reported from the Fitbit Charge 2.
Very Active Minutes | Length of stay in the inpatient facility-will differ for each patient (expected average of 3 weeks)
  Very active minutes will be reported from the Fitbit Charge 2.
Minutes Asleep | Length of stay in the inpatient facility-will differ for each patient (expected average of 3 weeks)
  Minutes asleep will be reported from the Fitbit Charge 2.

SECONDARY OUTCOMES:
Cognitive Function via the FIM Instrument | Length of stay in the inpatient facility-will differ for each patient (expected average of 3 weeks)
  The FIM® instrument (FIM) provides a uniform system of measurement for disability based on the International Classification of Impairment, Disabilities and Handicaps. It measures the level of a patient's disability and indicates how much assistance is required for the individual to carry out activities of daily living. The FIM contains 18 items composed of 13 motor tasks and 5 cognitive tasks (considered basic activities of daily living). Tasks are rated on a 7 point ordinal scale that ranges from total assistance (or complete dependence) to complete independence. Scores range from 18 (lowest) to 126 (highest) indicating level of function. Scores are generally rated at admission and discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Cooper, PT, DPT, NCS, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No